CLINICAL TRIAL: NCT01995838
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Bayesian Adaptive Randomization Design, Dose Response Study of the Efficacy of E2006 in Adults and Elderly Subjects With Chronic Insomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2006-G000-201
Record Dates: First submitted 2013-11-13; First posted 2013-11-27 (Estimated); Results first posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2015-11

CONDITIONS: Chronic Insomnia; Adults; Elderly
Keywords: Chronic Insomnia; Adults; Elderly
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- E2006 (Experimental): E2006 1 mg, 2.5 mg, 5 mg, 10 mg, 15 mg, or 25 mg, in tablet form, taken orally, 30 minutes prior to bedtime, each night for 15 consecutive nights
  Interventions: Drug: E2006
- Placebo (Placebo Comparator): E2006-matched placebo in tablet form, taken orally, 30 minutes prior to bedtime, each night for 15 consecutive nights
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E2006 — E2006 1 mg, 2.5 mg, 5 mg, 10 mg, 15 mg, or 25 mg, in tablet form, taken orally, 30 minutes prior to bedtime, each night for 15 consecutive nights
  Arms: E2006
Drug: Placebo — E2006-matched placebo in tablet form, taken orally, 30 minutes prior to bedtime, each night for 15 consecutive nights
  Arms: Placebo

SUMMARY:
This is a multicenter, multiple dose, randomized, double-blind, placebo-controlled, parallel-group, Bayesian adaptive, dose response study in subjects with chronic insomnia. Subjects will be randomized to 1 of 6 doses of E2006 (1 mg, 2.5 mg, 5 mg, 10 mg, 15 mg, or 25 mg) or placebo.

DETAILED DESCRIPTION:
The study will have 2 phases, Prerandomization and Randomization. The Prerandomization Phase will last up to 21 days and will consist of a Screening Period (Days -21 to -2) and a Baseline Period (Day -1). Following the Baseline Period, all eligible subjects will be randomized, in a double-blind manner, to receive E2006 or placebo for 15 nights during the Treatment Period (Days 1 to 15), then all subjects will receive placebo, in a single-blind manner, for 2 nights (Days 16 to 17) during the Rebound Insomnia Assessment Period (Days 16 to 18). Subjects will not receive any treatment during the Follow-up Period (Days 19 to 29). All subjects will come to the clinic for screening procedures. During the Screening Period, subjects will complete the Sleep Diary each day. Polysomnographic sleep will be measured during the Screening Period on 2 consecutive nights between Day -9 and Day -3. These 8-hour polysomnograms (PSGs) will start at the median habitual bedtime calculated from responses on the Sleep Diary completed 7 days immediately prior to the first PSG night. Subjects may leave the clinic between the screening/baseline PSG nights.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following criteria to be included in this study:

1. Male or female subjects age 18 to 80 years at the time of informed consent
2. Meets the 5th Edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for Insomnia Disorder
3. Subjective Sleep Onset Latency (sSOL) typically greater than or equal to 30 minutes in the last 4 weeks and/or subjective WASO (sWASO) typically greater than or equal to 60 minutes in the last 4 weeks
4. Regular time in bed between 6.5 and 9.0 hours
5. Regular bedtime between 21:00 and 24:00 and regular waketime between 05:00 and 09:00
6. Insomnia Severity Index (ISI) score greater than or equal to 15 at Screening
7. Confirmation of current insomnia symptoms as determined from responses on the Sleep Diary completed for 7 nights prior to the first screening/baseline PSG
8. Objective (PSG) evidence of insomnia at the screening/baseline PSGs as follows:

   1. LPS average greater than or equal to 30 minutes on the 2 consecutive screening/baseline PSGs, with neither night lesser than 15 minutes and/or
   2. WASO average greater than or equal to 30 minutes on the 2 consecutive screening/baseline PSGs, with neither night lesser than 20 minutes
   3. SE average lesser than or equal to 85% on the 2 consecutive screening/baseline PSGs, with neither night greater than 87.5%
9. Females of childbearing potential must not have had unprotected sexual intercourse within 30 days before study entry and must agree to use two highly effective method of contraception
10. Male subjects must have had a successful vasectomy (confirmed azoospermia) or they and their female partners must meet the criteria above (i.e., not of childbearing potential or practicing highly effective contraception throughout the study period and for 30 days after study drug discontinuation). No sperm donation is allowed during the study period and for 30 days after study drug discontinuation.
11. Provide written informed consent
12. Willing to stay in bed for at least 8 hours each night spent in the clinic
13. Willing and able to comply with all aspects of the protocol

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from this study:

1. Females who are pregnant (positive beta-human chorionic gonadotropin [B-hCG] test) or breastfeeding
2. Any lifetime diagnosis of sleep-related breathing disorder, periodic limb movement disorder, restless legs syndrome, nightmare disorder, sleep terror disorder, sleepwalking disorder, rapid eye movement (REM) behavior disorder, or narcolepsy
3. Aged 18 to 64 years: Apnea-Hypopnea Index greater than or equal to 10, or Periodic Limb Movements with Arousal Index greater than or equal to 10 on first (diagnostic) PSG night at Screening. Aged 65 to 80 years: Apnea-Hypopnea Index greater than 15, or Periodic Limb Movements with Arousal Index greater than 15 on first (diagnostic) PSG night at Screening
4. Beck Depression Inventory (BDI) - II score greater than 19 at Screening
5. Beck Anxiety Inventory (BAI) score greater than 15 at Screening
6. Used a prescription for any modality of treatment for insomnia, including cognitive behavioral therapy, within 2 weeks prior to screening/baseline PSG, or between Screening and Baseline
7. Used any medication or sleep aid with known effects on sleep, within 2 weeks prior to screening/baseline PSG, or between Screening and Baseline
8. Used any prohibited prescription or over-the-counter concomitant medications within the week prior to the first screening/baseline PSG.
9. Transmeridian travel across 3 or more time zones in the 2 weeks prior to Screening, or plans to travel across 3 or more time zones during study
10. Unwilling to limit caffeine consumption to lesser than or equal to 600 mg caffeine (approximately four 6-oz cups of caffeinated coffee, or three 12-oz caffeinated sodas, or three 8-oz caffeinated tea beverages), avoid caffeine after 18:00 throughout the study, and avoid caffeine after 13:00 on PSG visits
11. Unwilling to limit alcohol intake to two or fewer drinks per day throughout the study, or to refrain from any alcohol for 3 hours prior to bedtime while at home throughout the study, or any alcohol on days and nights spent in the clinic. A drink is defined as approximately 12 oz (360 mL) of beer, 4 oz (120 mL) of wine, or 1 oz (30 mL) of liquor.
12. Any subject that has a known history of malaria or has traveled to a country with known malarial risk (i.e., are designated as 'high' or 'moderate' risk country according to the list available at http://www.cdc.gov/malaria) within the last year.
13. A prolonged QT/QT interval corrected for heart rate (QTc) interval (QTc greater than 450 ms) as demonstrated by a repeated electrocardiogram (ECG) at Screening (repeated only if initial ECG indicates a QTc interval greater than 450 ms). A history of risk factors for torsade de pointes (e.g., heart failure, hypokalemia, family history of long QT Syndrome) or the use of concomitant medications that prolong the QT/QTc interval.
14. Any suicidal ideation with intent with or without a plan at Screening, Baseline, or within 6 months before Screening (i.e., answering "Yes" to questions 4 or 5 on the Suicidal Ideation section of the Columbia-Suicide Severity Rating Scale [C-SSRS])
15. Any lifetime suicidal behavior (per the Suicidal Behavior Section of the C-SSRS)
16. Evidence of clinically significant disease (e.g., cardiac, respiratory, gastrointestinal, renal disease) that in the opinion of the investigator(s) could affect the subject's safety or interfere with the study assessments
17. Hypersensitivity to the study drug or any of the excipients
18. Any history of a medical condition or a concomitant medical condition that in the opinion of the investigator(s) would compromise the subject's ability to safely complete the study
19. Scheduled for surgery during the study
20. Known to be human immunodeficiency virus (HIV) positive
21. Active viral hepatitis (B or C) as demonstrated by positive serology
22. Psychotic disorder(s) or unstable recurrent affective disorder(s) evident by use of antipsychotics or prior suicide attempt(s) within approximately the last 2 years
23. History of drug or alcohol dependency or abuse within approximately the last 2 years
24. Unwilling to refrain from use of illegal (or legalized) recreational drugs during the study or test positive for illegal (or legalized) drugs at Screening, Baseline, or Day 14
25. Currently enrolled in another clinical trial or used any investigational drug or device within 30 days or 5x the half-life, whichever is longer preceding informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2013-11-13 (Actual); Primary Completion 2014-04-29 (Actual); Study Completion 2014-04-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Glendale, Arizona
  - Phoenix, Arizona
  - Fountain Valley, California
  - Oceanside, California
  - San Diego, California
  - Thousand Oaks, California
  - Colorado Springs, Colorado
  - Brandon, Florida
  - Hallandale, Florida
  - Hollywood, Florida
  - South Miami, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Overland Park, Kansas
  - Glen Burnie, Maryland
  - Las Vegas, Nevada
  - New York, New York
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Columbia, South Carolina
  - Austin, Texas
  - Dallas, Texas
  - Vienna, Virginia

REFERENCES:
- [Derived] Murphy P, Moline M, Mayleben D, Rosenberg R, Zammit G, Pinner K, Dhadda S, Hong Q, Giorgi L, Satlin A. Lemborexant, A Dual Orexin Receptor Antagonist (DORA) for the Treatment of Insomnia Disorder: Results From a Bayesian, Adaptive, Randomized, Double-Blind, Placebo-Controlled Study. J Clin Sleep Med. 2017 Nov 15;13(11):1289-1299. doi: 10.5664/jcsm.6800. PMID 29065953

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 23 investigative sites in the United States from 13 Nov 2013 to 29 Apr 2014.
Pre-assignment Details: A total of 616 participants were screened, of which 325 were screen failures and 291 were randomized to receive study treatment.
Groups:
- Placebo: Participants received lemborexant placebo-matching tablets, orally, once daily on Day 1 to Day 15 in the double-blind treatment phase, followed by lemborexant placebo-matching tablets, orally, once daily on Days 16 and 17 in the single-blind placebo run-out phase.
- Lemborexant 1 Milligram (mg): Participants received lemborexant 1 mg tablets, orally, once daily on Day 1 to Day 15 in the double-blind treatment phase, followed by lemborexant placebo-matching tablets, orally, once on Days 16 and 17 in the single-blind placebo run-out phase.
- Lemborexant 2.5 mg: Participants received lemborexant 2.5 mg tablets, orally, once daily on Day 1 to Day 15 in the double-blind treatment phase, followed by lemborexant placebo-matching tablets, orally, once daily on Days 16 and 17 in the single-blind placebo run-out phase.
- Lemborexant 5 mg: Participants received lemborexant 5 mg tablets, orally, once daily on Day 1 to Day 15 in the double-blind treatment phase, followed by lemborexant placebo-matching tablets, orally, once daily on Days 16 and 17 in the single-blind placebo run-out phase.
- Lemborexant 10 mg: Participants received lemborexant 10 mg tablets, orally, once daily on Day 1 to Day 15 in the double-blind treatment phase, followed by lemborexant placebo-matching tablets, orally, once daily on Days 16 and 17 in the single-blind placebo run-out phase.
- Lemborexant 15 mg: Participants received lemborexant 15 mg tablets, orally, once daily on Day 1 to Day 15 in the double-blind treatment phase, followed by lemborexant placebo-matching tablets, orally, once daily on Days 16 and 17 in the single-blind placebo run-out phase.
- Lemborexant 25 mg: Participants received lemborexant 25 mg tablets, orally, once daily on Day 1 to Day 15 in the double-blind treatment phase, followed by lemborexant placebo-matching tablets, orally, once daily on Days 16 and 17 in the single-blind placebo run-out phase.
Period: Overall Study
Arm/Group | Placebo | Lemborexant 1 Milligram (mg) | Lemborexant 2.5 mg | Lemborexant 5 mg | Lemborexant 10 mg | Lemborexant 15 mg | Lemborexant 25 mg
Started | 56 | 32 | 27 | 38 | 32 | 56 | 50
Completed | 51 | 30 | 27 | 36 | 30 | 54 | 45
Not Completed | 5 | 2 | 0 | 2 | 2 | 2 | 5
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Participant choice | 2 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other | 3 | 1 | 0 | 2 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least 1 dose of study drug and had at least 1 postdose safety assessment.
Groups:
- Lemborexant 1 mg: Participants received lemborexant 1 mg tablets, orally, once daily on Day 1 to Day 15 in the double-blind treatment phase, followed by lemborexant placebo-matching tablets, orally, once on Days 16 and 17 in the single-blind placebo run-out phase.
- Total: Total of all reporting groups
Arm/Group | Lemborexant 1 mg | Lemborexant 2.5 mg | Lemborexant 5 mg | Lemborexant 10 mg | Lemborexant 15 mg | Lemborexant 25 mg | Placebo | Total
Number analyzed (Participants) | 32 | 27 | 38 | 32 | 56 | 50 | 56 | 291
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.3 (13.0) | 49.7 (14.3) | 51.1 (14.3) | 47.1 (13.7) | 44.0 (14.6) | 48.9 (13.4) | 47.1 (15.6) | 48.3 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 17 | 23 | 20 | 32 | 31 | 36 | 182
  Male | 9 | 10 | 15 | 12 | 24 | 19 | 20 | 109

OUTCOME MEASURES:

1. Primary Outcome: Probability of Having Utility Function Greater Than (>) 1 Based on Bayesian Analysis
Description: The utility of a dose was a function of both Sleep Efficiency (SE) and Karolinska Sleepiness Scale (KSS), constructed by specifying the 1-dimensional component for each outcome measure and then combining them multiplicatively. Sufficient utility was defined as a probability of having utility function >1. Probability of having utility function >1 at the end of study visit (full analysis) was reported.
Time Frame: Baseline up to Day 3
Population: The full analysis set (FAS) included all participants who were randomized, received at least 1 dose of study drug and had at least 1 postdose primary efficacy measurement.
Measure: Number; unit: probability
Arm/Group | Lemborexant 1 mg | Lemborexant 2.5 mg | Lemborexant 5 mg | Lemborexant 10 mg | Lemborexant 15 mg | Lemborexant 25 mg
Number analyzed (Participants) | 32 | 27 | 38 | 32 | 56 | 50
probability | 0.8789 | 0.8920 | 0.9032 | 0.9406 | 0.9866 | 0.9675

2. Primary Outcome: Mean Change From Baseline in Karolinska Sleepiness Scale (KSS) Score at End of Treatment
Description: The KSS was used to measure next-day residual effects at prespecified time points. The KSS was a 9-point scale on which the participant rated their sleepiness from 1 (extremely alert) to 9 (extremely sleepy/fighting sleep), where higher scores indicated an increase in sleepiness. The end of treatment score was calculated by the mean scores at the timepoint at 1 hour after morning wake time of Day 15 and 16.
Time Frame: 1 hour after morning wake time at Baseline and Days 15-16
Population: The FAS included all participants who were randomized, received at least 1 dose of study drug and had at least 1 post-dose primary efficacy measurement. Here, number of participants analyzed (N) represents participants who were available for analysis at the specified timepoints.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Lemborexant 1 mg | Lemborexant 2.5 mg | Lemborexant 5 mg | Lemborexant 10 mg | Lemborexant 15 mg | Lemborexant 25 mg | Placebo
Number analyzed (Participants) | 31 | 27 | 37 | 31 | 54 | 46 | 51
Units on a scale | 0.29 (0.219) | -0.10 (0.234) | 0.20 (0.200) | -0.22 (0.219) | 0.16 (0.166) | 0.45 (0.180) | -0.23 (0.170)
Statistical Analysis 1: Comparison: Lemborexant 1 mg vs Placebo; Test type: Superiority; p = 0.0651, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = 0.51, 95% CI 2-sided [-0.03 to 1.06]
Statistical Analysis 2: Comparison: Lemborexant 2.5 mg vs Placebo; Test type: Superiority; p = 0.6490, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = 0.13, 95% CI 2-sided [-0.44 to 0.70]
Statistical Analysis 3: Comparison: Lemborexant 5 mg vs Placebo; Test type: Superiority; p = 0.1059, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = 0.43, 95% CI 2-sided [-0.09 to 0.94]
Statistical Analysis 4: Comparison: Lemborexant 10 mg vs Placebo; Test type: Superiority; p = 0. 9818, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = 0.01, 95% CI 2-sided [-0. 54 to 0.55]
Statistical Analysis 5: Comparison: Lemborexant 15 mg vs Placebo; Test type: Superiority; p = 0. 1071, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = 0.38, 95% CI 2-sided [-0.08 to 0.85]
Statistical Analysis 6: Comparison: Lemborexant 25 mg vs Placebo; Test type: Superiority; p = 0.0063, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = 0.68, 95% CI 2-sided [0.19 to 1.17]

3. Secondary Outcome: Mean Change From Baseline in Sleep Efficiency (SE) After Dosing on Days 1-2 and Days 14-15
Description: Sleep efficiency was calculated as total sleep time divided by time spent in bed multiplied by 100. An increase in SE indicated improvement in sleeping, such that, the participant spends more time in bed asleep. Mean scores of Days 1-2 and Days 14-15 were used to evaluate change from baseline.
Time Frame: Baseline, Days 1-2, and Days 14-15
Population: The FAS included all participants who were randomized, received at least 1 dose of study drug, had at least 1 post-dose primary efficacy measurement with both baseline and post baseline data available for analysis at each timepoints.
Measure: Least Squares Mean (Standard Error); unit: percentage of sleep time
Arm/Group | Lemborexant 1 mg | Lemborexant 2.5 mg | Lemborexant 5 mg | Lemborexant 10 mg | Lemborexant 15 mg | Lemborexant 25 mg | Placebo
Number analyzed (Participants) | 32 | 27 | 38 | 32 | 56 | 50 | 56
percentage of sleep time
  Days 1-2 | 18.72 (1.366) | 18.59 (1.487) | 19.89 (1.250) | 22.25 (1.361) | 24.22 (1.029) | 24.28 (1.091) | 14.16 (1.031)
  Days 14-15 | 14.43 (1.428) | 18.02 (1.528) | 19.85 (1.302) | 21.87 (1.421) | 21.97 (1.077) | 22.96 (1.169) | 14.08 (1.100)
Statistical Analysis 1: Comparison: Lemborexant 1 mg vs Placebo; Days 1-2; Test type: Superiority; p = 0.0083, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = 4.57, 95% CI 2-sided [1.19 to 7.94]
Statistical Analysis 2: Comparison: Lemborexant 2.5 mg vs Placebo; Days 1-2; Test type: Superiority; p = 0.0151, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = 4.44, 95% CI 2-sided [0.86 to 8.01]
Statistical Analysis 3: Comparison: Lemborexant 5 mg vs Placebo; Days 1-2; Test type: Superiority; p = 0.0005, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = 5.74, 95% CI 2-sided [2.54 to 8.93]
Statistical Analysis 4: Comparison: Lemborexant 10 mg vs Placebo; Days 1-2; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = 8.09, 95% CI 2-sided [4.73 to 11.45]
Statistical Analysis 5: Comparison: Lemborexant 15 mg vs Placebo; Days 1-2; Test type: Superiority; p < 0.0001, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = 10.06, 95% CI 2-sided [7.20 to 12.93]
Statistical Analysis 6: Comparison: Lemborexant 25 mg vs Placebo; Days 1-2; Test type: Superiority; p < 0.0001, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = 10.13, 95% CI 2-sided [7.18 to 13.08]
Statistical Analysis 7: Comparison: Lemborexant 1 mg vs Placebo; Days 14-15; Test type: Superiority; p = 0.8505, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = 0.34, 95% CI 2-sided [-3.22 to 3.90]
Statistical Analysis 8: Comparison: Lemborexant 2.5 mg vs Placebo; Days 14-15; Test type: Superiority; p = 0.0380, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = 3.94, 95% CI 2-sided [0.22 to 7.66]
Statistical Analysis 9: Comparison: Lemborexant 5 mg vs Placebo; Days 14-15; Test type: Superiority; p = 0.0008, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = 5.76, 95% CI 2-sided [2.40 to 9.12]
Statistical Analysis 10: Comparison: Lemborexant 10 mg vs Placebo; Days 14-15; Test type: Superiority; p < 0.0001, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = 7.78, 95% CI 2-sided [4.24 to 11.32]
Statistical Analysis 11: Comparison: Lemborexant 15 mg vs Placebo; Days 14-15; Test type: Superiority; p < 0.0001, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = 7.89, 95% CI 2-sided [4.86 to 10.92]
Statistical Analysis 12: Comparison: Lemborexant 25 mg vs Placebo; Days 14-15; Test type: Superiority; p < 0.0001, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = 8.87, 95% CI 2-sided [5.72 to 12.02]

4. Secondary Outcome: Mean Change From Baseline in Latency to Persistent Sleep (LPS) After Dosing on Days 1-2 and Days 14-15
Description: LPS was calculated as minutes from lights off to the first 30-second epoch of 20 consecutive epochs of non-wakefulness. A decrease in LPS indicated improvement in time needed to fall asleep. Mean scores of Days 1-2 and Days 14-15 were used to evaluate change from baseline.
Time Frame: Baseline, Days 1-2, and Days 14-15
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Lemborexant 1 mg | Lemborexant 2.5 mg | Lemborexant 5 mg | Lemborexant 10 mg | Lemborexant 15 mg | Lemborexant 25 mg | Placebo
Number analyzed (Participants) | 32 | 27 | 38 | 32 | 56 | 50 | 56
minutes
  Days 1-2 | -42.92 (41.855) | -52.74 (50.149) | -47.72 (39.389) | -46.80 (46.106) | -51.59 (36.728) | -50.16 (43.140) | -22.90 (44.457)
  Days 14-15 | -41.23 (34.618) | -54.24 (44.918) | -51.86 (41.994) | -56.14 (45.553) | -51.95 (41.926) | -50.79 (40.160) | -22.43 (29.045)
Statistical Analysis 1: Comparison: Lemborexant 1 mg vs Placebo; Days 1-2; Test type: Superiority; p = 0.1407, ANCOVA; Baseline value and treatment as covariates; Geometric Mean Ratio = 0.77, 95% CI 2-sided [0.54 to 1.09]
Statistical Analysis 2: Comparison: Lemborexant 2.5 mg vs Placebo; Test type: Superiority — Days 1-2; p = 0.0018, ANCOVA; Baseline value and treatment as covariates; Geometric Mean Ratio = 0.55, 95% CI 2-sided [0.38 to 0.80]
Statistical Analysis 3: Comparison: Lemborexant 5 mg vs Placebo; Days 1-2; Test type: Superiority; p = 0.0025, ANCOVA; Baseline value and treatment as covariates; Geometric Mean Ratio = 0.60, 95% CI 2-sided [0.43 to 0.83]
Statistical Analysis 4: Comparison: Lemborexant 10 mg vs Placebo; Days 1-2; Test type: Superiority; p = 0.0006, ANCOVA; Baseline value and treatment as covariates; Geometric Mean Ratio = 0.54, 95% CI 2-sided [0.38 to 0.76]
Statistical Analysis 5: Comparison: Lemborexant 15 mg vs Placebo; Days 1-2; Test type: Superiority; p < 0.0001, ANCOVA; Baseline value and treatment as covariates; Geometric Mean Ratio = 0.52, 95% CI 2-sided [0.38 to 0.70]
Statistical Analysis 6: Comparison: Lemborexant 25 mg vs Placebo; Days 1-2:; Test type: Superiority; p < 0.0001, ANCOVA; Baseline value and treatment as covariates; Geometric Mean Ratio = 0.39, 95% CI 2-sided [0.29 to 0.54]
Statistical Analysis 7: Comparison: Lemborexant 1 mg vs Placebo; Days 14-15; Test type: Superiority; p = 0.1158, ANCOVA; Baseline value and treatment as covariates; Geometric Mean Ratio = 0.73, 95% CI 2-sided [0.49 to 1.08]
Statistical Analysis 8: Comparison: Lemborexant 2.5 mg vs Placebo; Days 14-15; Test type: Superiority; p = 0.0010, ANCOVA; Baseline value and treatment as covariates; Geometric Mean Ratio = 0.49, 95% CI 2-sided [0.33 to 0.75]
Statistical Analysis 9: Comparison: Lemborexant 5 mg vs Placebo; Days 14-15; Test type: Superiority; p < 0.0001, ANCOVA; Baseline value and treatment as covariates; Geometric Mean Ratio = 0.47, 95% CI 2-sided [0.32 to 0.69]
Statistical Analysis 10: Comparison: Lemborexant 10 mg vs Placebo; Days 14-15; Test type: Superiority; p < 0.0001, ANCOVA; Baseline value and treatment as covariates; Geometric Mean Ratio = 0.32, 95% CI 2-sided [0.21 to 0.47]
Statistical Analysis 11: Comparison: Lemborexant 15 mg vs Placebo; Days 14-15; Test type: Superiority; p < 0.0001, ANCOVA; Baseline value and treatment as covariates; Geometric Mean Ratio = 0.41, 95% CI 2-sided [0.29 to 0.57]
Statistical Analysis 12: Comparison: Lemborexant 25 mg vs Placebo; Days 14-15; Test type: Superiority; p < 0.0001, ANCOVA; Baseline value and treatment as covariates; Geometric Mean Ratio = 0.34, 95% CI 2-sided [0.24 to 0.48]

5. Secondary Outcome: Mean Change From Baseline in Wakefulness After Sleep Onset (WASO) After Dosing on Days 1-2 and Days 14-15
Description: WASO was calculated as minutes of wakefulness from the onset of persistent sleep until lights on. A decrease in WASO indicated improvement in sleep maintenance. Mean scores of Days 1-2 and Days 14-15 were used to evaluate change from baseline.
Time Frame: Baseline, Days 1-2, and Days 14-15
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Lemborexant 1 mg | Lemborexant 2.5 mg | Lemborexant 5 mg | Lemborexant 10 mg | Lemborexant 15 mg | Lemborexant 25 mg | Placebo
Number analyzed (Participants) | 32 | 27 | 38 | 32 | 56 | 50 | 56
minutes
  Days 1-2 | -52.11 (5.441) | -43.33 (5.915) | -52.29 (5.423) | -60.84 (1.302) | -70.38 (4.103) | -66.87 (4.342) | -41.03 (4.095)
  Days 14-15: number analyzed (Participants) | 31 | 27 | 37 | 31 | 54 | 46 | 52
  Days 14-15 | -32.46 (6.159) | -40.47 (6.581) | -48.84 (5.609) | -52.88 (6.129) | -58.95 (4.651) | -59.67 (5.039) | -38.15 (4.728)
Statistical Analysis 1: Comparison: Lemborexant 1 mg vs Placebo; Days 1-2; Test type: Superiority; p = 0.1050, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = -11.08, 95% CI 2-sided [-24.48 to 2.33]
Statistical Analysis 2: Comparison: Lemborexant 2.5 mg vs Placebo; Days 1-2; Test type: Superiority; p = 0.7501, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = -2.29, 95% CI 2-sided [-16.46 to 11.87]
Statistical Analysis 3: Comparison: Lemborexant 5 mg vs Placebo; Days 1-2; Test type: Superiority; p = 0.0818, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = -11.26, 95% CI 2-sided [-23.94 to 1.43]
Statistical Analysis 4: Comparison: Lemborexant 10 mg vs Placebo; Days 1-2; Test type: Superiority; p = 0.0038, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = -19.81, 95% CI 2-sided [-33.18 to -6.43]
Statistical Analysis 5: Comparison: Lemborexant 15 mg vs Placebo; Days 1-2; Test type: Superiority; p < 0.0001, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = -29.34, 95% CI 2-sided [-40.75 to 17.93]
Statistical Analysis 6: Comparison: Lemborexant 25 mg vs Placebo; Days 1-2; Test type: Superiority; p < 0.0001, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = -25.84, 95% CI 2-sided [-37.59 to -14.09]
Statistical Analysis 7: Comparison: Lemborexant 1 mg vs Placebo; Days 14-15; Test type: Superiority; p = 0.4642, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = 0.4642, 95% CI 2-sided [-9.60 to 20.98]
Statistical Analysis 8: Comparison: Lemborexant 2.5 mg vs Placebo; Days 14-15; Test type: Superiority — Baseline value and treatment as covariates; p = 0.7754, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = -2.31, 95% CI 2-sided [-18.27 to 13.64]
Statistical Analysis 9: Comparison: Lemborexant 5 mg vs Placebo; Days 14-15; Test type: Superiority; p = 0.1461, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = -10.69, 95% CI 2-sided [-25.14 to 3.75]
Statistical Analysis 10: Comparison: Lemborexant 10 mg vs Placebo; Days 14-15; Test type: Superiority; p = 0.0581, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = -14.73, 95% CI 2-sided [-29.97 to 0.51]
Statistical Analysis 11: Comparison: Lemborexant 15 mg vs Placebo; Days 14-15; Test type: Superiority; p = 0.0019, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = -20.80, 95% CI 2-sided [-33.86 to -7.74]
Statistical Analysis 12: Comparison: Lemborexant 25 mg vs Placebo; Days 14-15; Test type: Superiority; p = 0.0020, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = -21.52, 95% CI 2-sided [-35.12 to -7.91]

6. Secondary Outcome: Potential Habituation Effect: Comparison Between Mean Change From Baseline in SE on Days 1-2 and Mean Change From Baseline in SE on Days 14-15
Description: Potential habituation effect evaluated the possibility of participants being habituated to changes in sleep during the 15 days of treatment with lemborexant. Data reported here was calculated as change from baseline of mean SE of Days 14-15 minus change from baseline of mean SE of Days 1-2. An increase in SE indicated improvement in sleeping, such that, the participant spends more time in bed asleep.
Time Frame: Baseline, Days 1-2, and Days 14-15
Population: The FAS included all participants who were randomized, received at least 1 dose of study drug and had at least 1 post-dose primary efficacy measurement. Here, overall number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of sleep time
Arm/Group | Lemborexant 1 mg | Lemborexant 2.5 mg | Lemborexant 5 mg | Lemborexant 10 mg | Lemborexant 15 mg | Lemborexant 25 mg | Placebo
Number analyzed (Participants) | 31 | 27 | 37 | 31 | 54 | 46 | 52
percentage of sleep time | -4.04 (8.194) | -0.54 (10.505) | 0.06 (6.888) | -0.68 (6.883) | -2.33 (6.600) | -2.15 (5.388) | -1.05 (7.192)

7. Secondary Outcome: Potential Habituation Effect: Comparison Between Mean Change From Baseline in Latency to Persistent Sleep (LPS) on Days 1-2 and Mean Change From Baseline in LPS on Days 14-15
Description: Potential habituation effect evaluated the possibility of participants being habituated to changes in sleep during the 15 days of treatment with lemborexant. Data reported here was calculated as change from baseline of mean LPS of Days 14-15 minus change from baseline of mean LPS of Days 1-2. LPS was calculated as minutes from lights off to the first 30-second epoch of 20 consecutive epochs of non-wakefulness. A decrease in LPS indicated improvement in time needed to fall asleep.
Time Frame: Baseline and Days 1-2, and Days 14-15
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Placebo: Days 1 to 15: Three E2006-matched placebo tablets were taken orally, 30 minutes before bedtime, each night for 15 consecutive nights. Days 16 to 18: Two E2006-matched placebo tablets were taken for 2 consecutive nights. Days 10 to 30: No study drug, E2006 or placebo, was taken.
Arm/Group | Lemborexant 1 mg | Lemborexant 2.5 mg | Lemborexant 5 mg | Lemborexant 10 mg | Lemborexant 15 mg | Lemborexant 25 mg | Placebo
Number analyzed (Participants) | 31 | 27 | 37 | 31 | 54 | 46 | 52
minutes | 2.71 (24.333) | -1.50 (22.120) | -4.60 (22.337) | -7.93 (17.415) | -1.11 (24.568) | 1.38 (12.046) | 0.57 (40.855)

8. Secondary Outcome: Potential Habituation Effect: Comparison Between Mean Change From Baseline in Wakefulness After Sleep Onset (WASO) on Days 1-2 and Mean Change From Baseline in WASO on Days 14-15
Description: Potential habituation effect evaluated the possibility of participants being habituated to changes in sleep during the 15 days of treatment with lemborexant. Data reported here was calculated as change from baseline of mean WASO of Days 14-15 minus change from baseline of mean WASO of Days 1-2. WASO was calculated as minutes of wakefulness from the onset of persistent sleep until lights on. A decrease in WASO indicated improvement in sleep maintenance.
Time Frame: Baseline, Days 1-2, and Days 14-15
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Lemborexant 1 mg | Lemborexant 2.5 mg | Lemborexant 5 mg | Lemborexant 10 mg | Lemborexant 15 mg | Lemborexant 25 mg | Placebo
Number analyzed (Participants) | 31 | 27 | 36 | 31 | 54 | 45 | 52
minutes | 17.98 (34.299) | 2.16 (44.054) | 2.68 (29.726) | 9.30 (25.890) | 11.76 (26.187) | 9.28 (23.119) | 5.99 (31.417)

9. Secondary Outcome: Rebound Insomnia: Mean Change From Baseline in Sleep Efficiency (SE) After Dosing on Days 16-17
Description: Rebound insomnia was assessed by comparing the change from baseline of the mean SE on Days 16-17. Sleep efficiency was calculated as total sleep time divided by time spent in bed multiplied by 100. An increase in SE indicated improvement in sleeping, such that, the participant spends more time in bed asleep. A negative change from baseline in SE indicated that SE was worse on Days 16 and 17 than at Baseline, which was considered as evidence for rebound insomnia.
Time Frame: Baseline and Days 16-17
Population: The FAS included all participants who were randomized, received at least 1 dose of study drug and had at least 1 post-dose primary efficacy measurement. Here, number of participants analyzed (N) represents participants who were available for analysis at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: percentage of sleep time
Arm/Group | Lemborexant 1 mg | Lemborexant 2.5 mg | Lemborexant 5 mg | Lemborexant 10 mg | Lemborexant 15 mg | Lemborexant 25 mg | Placebo
Number analyzed (Participants) | 31 | 27 | 36 | 31 | 54 | 45 | 52
percentage of sleep time | 13.12 (1.661) | 15.53 (1.777) | 17.67 (1.535) | 13.78 (1.653) | 18.58 (1.253) | 17.12 (1.374) | 16.17 (1.280)
Statistical Analysis 1: Comparison: Lemborexant 1 mg vs Placebo; Days 16-17; Test type: Superiority; p = 0.1483, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = -3.05, 95% CI 2-sided [-7.20 to 1.09]
Statistical Analysis 2: Comparison: Lemborexant 2.5 mg vs Placebo; Days 16-17; Test type: Superiority; p = 0.7720, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = -0.64, 95% CI 2-sided [-4.96 to 3.69]
Statistical Analysis 3: Comparison: Lemborexant 5 mg vs Placebo; Days 16-17; Test type: Superiority; p = 0.4548, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = 1.50, 95% CI 2-sided [-2.44 to 5.44]
Statistical Analysis 4: Comparison: Lemborexant 10 mg vs Placebo; Days 16-17; Test type: Superiority; p = 0.2530, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = -2.39, 95% CI 2-sided [-6.51 to 1.72]
Statistical Analysis 5: Comparison: Lemborexant 15 mg vs Placebo; Days 16-17; Test type: Superiority; p = 0.1794, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = 2.41, 95% CI 2-sided [-1.11 to 5.93]
Statistical Analysis 6: Comparison: Lemborexant 25 mg vs Placebo; Days 16-17; Test type: Superiority; p = 0.6148, ANCOVA; Baseline value and treatment as covariates; LS Mean Difference = 0.94, 95% CI 2-sided [-2.74 to 4.63]

10. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Event (TEAE) and Serious Adverse Event (SAE)
Time Frame: TEAEs: Baseline up to Day 30, SAEs: Baseline up to 30 days after last dose of study drug (up to 47 days)
Population: The safety analysis set included all participants who received at least 1 dose of study drug and had at least 1 post-dose safety assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Lemborexant 1 mg | Lemborexant 2.5 mg | Lemborexant 5 mg | Lemborexant 10 mg | Lemborexant 15 mg | Lemborexant 25 mg | Placebo
Number analyzed (Participants) | 32 | 27 | 38 | 32 | 56 | 50 | 56
percentage of participants
  TEAE | 34.4 | 40.7 | 42.1 | 59.4 | 55.4 | 60.0 | 37.5
  SAE | 0 | 0 | 0 | 0 | 0 | 2.0 | 1.8

11. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Clinical Laboratory Parameters
Time Frame: Baseline up to Day 30
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Lemborexant 1 mg | Lemborexant 2.5 mg | Lemborexant 5 mg | Lemborexant 10 mg | Lemborexant 15 mg | Lemborexant 25 mg | Placebo
Number analyzed (Participants) | 32 | 27 | 38 | 32 | 56 | 50 | 56
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Time Frame: Baseline up to Day 30
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Lemborexant 1 mg | Lemborexant 2.5 mg | Lemborexant 5 mg | Lemborexant 10 mg | Lemborexant 15 mg | Lemborexant 25 mg | Placebo
Number analyzed (Participants) | 32 | 27 | 38 | 32 | 56 | 50 | 56
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Electrocardiogram (ECGs)
Time Frame: Baseline up to Day 30
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Lemborexant 1 mg | Lemborexant 2.5 mg | Lemborexant 5 mg | Lemborexant 10 mg | Lemborexant 15 mg | Lemborexant 25 mg | Placebo
Number analyzed (Participants) | 32 | 27 | 38 | 32 | 56 | 50 | 56
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: TEAEs: Baseline up to Day 30, SAEs: Baseline up to 30 days after last dose of study drug (up to 47 days)
Description: Safety analysis set included participants who received at least one dose of study drug and had at least one postdose safety assessment.
Arm/Group | Lemborexant 1 mg | Lemborexant 2.5 mg | Lemborexant 5 mg | Lemborexant 10 mg | Lemborexant 15 mg | Lemborexant 25 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/27 | 0/38 | 0/32 | 0/56 | 0/50 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/27 | 0/38 | 0/32 | 0/56 | 1/50 | 1/56
Other Adverse Events (participants affected / at risk) | 11/32 | 11/27 | 16/38 | 19/32 | 31/56 | 30/50 | 21/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lemborexant 1 mg (N=32) | Lemborexant 2.5 mg (N=27) | Lemborexant 5 mg (N=38) | Lemborexant 10 mg (N=32) | Lemborexant 15 mg (N=56) | Lemborexant 25 mg (N=50) | Placebo (N=56)
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Grand Mal Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lemborexant 1 mg (N=32) | Lemborexant 2.5 mg (N=27) | Lemborexant 5 mg (N=38) | Lemborexant 10 mg (N=32) | Lemborexant 15 mg (N=56) | Lemborexant 25 mg (N=50) | Placebo (N=56)
Somnolence (Nervous system disorders) | 1 | 1 | 2 | 4 | 10 | 11 | 0
Headache (Nervous system disorders) | 3 | 3 | 3 | 3 | 6 | 5 | 3
Sleep paralysis (Nervous system disorders) | 0 | 0 | 1 | 3 | 4 | 2 | 0
Rapid eye movements sleep abnormal (Psychiatric disorders) | 0 | 2 | 1 | 1 | 3 | 2 | 2
Nightmare (Psychiatric disorders) | 0 | 0 | 1 | 3 | 4 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 2 | 0 | 1 | 3 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 2 | 0 | 2 | 1 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 2 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 3 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cataplexy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sedation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sleep phase rhythm disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypnagogic hallucination (Psychiatric disorders) | 0 | 0 | 1 | 1 | 2 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 1
Elevated mood (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Anger (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bruxism (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Euphoric mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypervigilance (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sleep talking (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 1 | 1 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Feeling drunk (General disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Application site dermatitis (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Energy increased (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Irritability (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Application site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Abnormal sensation in eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Excessive eye blinking (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperacusis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diaphragmatic disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No